CLINICAL TRIAL: NCT03741699
Title: A Phase III Multicentre, Randomized, Unblinded Clinical Trial to Test the Effect of Treatment with Recombinant LH Prior to Controlled Ovarian Stimulation in Poor Ovarian Responder Women with an Advanced Maternal Age
Brief Title: Recombinant LH Prior to Ovarian Stimulation in Poor Ovarian Responders (PRE-LH)
Acronym: PRE-LH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Collaborators: Merck, S.L., Spain (Industry); Syntax for Science, S.L (Industry); Fundación IVI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601-ALC-002-MM; 2017-004298-15 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Infertility, Female
Keywords: Poor ovarian response; Recombinant LH; Advanced maternal age; Oocyte retrieved
MeSH Terms: conditions — Infertility, Female | interventions — Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Intervention Model Description: prospective, interventional, randomised, unblinded and controlled study with 2 parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - experimental group (Experimental): Treatment with 150 IU/day rLH, administered subcutaneously for 4 consecutive days prior to COS (with a starting dose of 225 IU/day rFSH and 75 IU/day rLH for 18 days maximum in a short antagonist protocol).
  Interventions: Drug: Pre-treatment with rLH (Luveris 75 IU),
- Arm 2 - control (no pre-treatment) group (No Intervention): The subjects assigned to this group will not receive any treatment in the four days prior to COS (with a starting dose of 225 IU/day rFSH and 75 IU/day rLH for 18 days maximum in a short antagonist protocol).

INTERVENTIONS:
Drug: Pre-treatment with rLH (Luveris 75 IU), — Treatment with 150 IU/day rLH (Luveris 75 IU), administered subcutaneously for 4 consecutive days prior to COS (Controlled ovarian stimulation)
  Arms: Arm 1 - experimental group

SUMMARY:
Controlled ovarian stimulation (COS) is one of the first stages of assisted reproductive treatment. The goal is to mimic the ovarian cycle while stimulating the ovaries to overproduce eggs capable of being fertilized, thus maximizing the chances of reproductive success. The stimulation phase involves the use of different hormonal medications but requires tests to check the development of follicles, and hormonal adjustment to get the optimal ovarian response to stimulation.

However, between 9 to 24% of patients fail to respond adequately to standard stimulation protocols, resulting in Poor Ovarian Response (POR). In addition to the low oocyte production, POR results in a restricted number of good quality embryos with appropriate implantation potential, suggesting a compromised oocyte quality.

POR is one of the most challenging problems in reproductive medicine. Poor responders are difficult to treat since their response to stimulation tend to be deficient even when using different drugs or protocols. In recent years, different therapeutic alternatives have been proposed for these patients. However, to date, the optimal stimulation protocol has not yet been described and oocyte donation is often offered as their only option to achieve pregnancy.

Recently, evidence has emerged that supplementation with a specific hormone, luteinizing hormone (LH), during or prior to COS could lead to improved reproductive outcomes in poor responders by increasing the number of oocytes retrieved and improving their quality.

The present study aims to evaluate the effect of the treatment with LH prior to COS on the ovarian response in patients with POR and advanced maternal age, the worst prognosis but more frequent group of poor responders attending fertility clinics. We will assess whether LH treatment prior to COS increases the number and quality of oocytes retrieved in those patients and, finally, analyse the impact in their chances of getting pregnant and having a baby.

ELIGIBILITY:
Inclusion Criteria:

1. -Patients with POR according to specific criteria that are in line with the criteria defined by the ESHRE (Bologna Criteria), according to which a patient is classified as a poor ovarian responder when she meets two of the three of the following criteria: I.- Previous episode of POR (≤3 oocytes) with conventional stimulation protocol II.- Abnormal ovarian reserve test with an antral follicle count (AFC) <5-7 and/or anti-mullerian hormone values (AMH) <0.5-1.1 ng/mL.

   III.- Women ≥40 years old and/or who have any other risk factor for POR. In addition, two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ovarian reserve test.
2. - Women ≥35 to ≤43 years for COS and assisted reproduction techniques (ART).
3. - Couple or single woman, accepting preimplantation genetic diagnosis (PGS) after blastocyst biopsy and delayed transfer for selection of euploid embryos.
4. - Body Mass Index (BMI) between18 and 30 kg/m 2 , inclusive.
5. - Ejaculatory sperm with concentration ≥ 5 mill spermatozoa/mL and ≥ 5 mill total spermatozoa progressive motility. Bank and cryopreserved semen allowed.
6. - Informed consent completed, signed and dated.

Exclusion Criteria:

1. - Cases of recurrent spontaneous miscarriage (≥2 clinical miscarriages) or implantation failure (after transfer of 6 good D3 embryos or 4 good blastocysts) will be excluded.
2. - Use of testicular or epididymal spermatozoa as well as ejaculate with concentration < 5 mill spermatozoa/mL and < 5 mill total spermatozoa progressive motility.
3. - Primary ovarian failure, PCOS (in accordance with the Rotterdam criteria) or ovary/s inaccessible for oocyte retrieval.
4. - Anatomical uterine abnormalities and any endometrium or myometrium pathology (adenomyosis, polyps, myoma, etc.) that may interfere with implantation or pregnancy. Patients with previous polypectomy, myomectomy or surgery for septate/subseptate/arcuatus uterus should not be excluded.
5. - Presence of unilateral or bilateral hydrosalpinx that has not been surgically removed or ligated.
6. - Presence of level III-IV endometriosis.
7. - History of tumours in the hypothalamus or pituitary gland, or ovarian, uterine or breast cancer.
8. - Abnormal bleeding of undetermined origin.
9. - Known infection with human immunodeficiency virus, active hepatitis B or C virus in the woman or her partner.
10. - Known allergy or hypersensitivity to the drugs administered during the trial.
11. - Concurrent significant medical pathologies that would endanger the patient's safety (uncontrolled thyroid or adrenal dysfunction, severe hepatic or renal impairment, etc.) or interfere with the test evaluations or the clinical outcomes (i.e. confirmed thrombophilia).
12. - Use of concomitant medication or any other circumstances that, in the opinion of the investigator, interferes with the development of the trial or does not ensure the safety and efficacy of the data.
13. - Simultaneous participation in another clinical trial or previous participation in this study.
14. - Participation in another clinical study two months before inclusion in the present study that could affect its objectives.

Ages: 35 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females
Enrollment: 88 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
number of oocytes retrieved | 37 days
  number of oocytes retrieved

SECONDARY OUTCOMES:
Number of follicles >17 mm on the previous day or the day of GnRH agonist injection (Decapeptyl) | from day 8-12 to day 33-37
P 4 and E 2 levels on the previous day or the day of GnRH agonist injection | from day 8-12 to day 33-37
Duration of stimulation and total gonadotropin dose during COS | from day 8-12 to day 33-37
Serum hormonal profile before and after IMP treatment and after stimulation | from day 8-12 to day 33-37
Cycle cancellation rates (stimulation cycle cancelled prior to oocyte retrieval if there is no follicular response after 10 days of stimulation or due to premature ovulation at any time before oocyte retrieval) | from day 8-12 to day 33-37
Number of mature or metaphase II (MII) oocytes/number of oocytes retrieved per puncture | Day 37
Number of retrieved oocytes/number of expected oocytes (follicles >15 mm on the day of GnRH agonist injection) | Day 37
Fertilization rate | Day 38
Hormonal profile in follicular fluid on the day of the puncture | Day 37
Gene expression profile in granulosa cells | Day 37
Apoptosis rate in granulosa cells | Day 37
Morphological variables of embryonic quality | Day 38 to 43
Blastocyst rate | Day 43
Number of optimal embryos (type A or B, according to ASEBIR classification) | Day 43
Number of euploid and aneuploid embryos | Day 50
Stimulation cycle yield (number of frozen embryos). | Day 43
Number of cycles with embryo transferred/ number of stimulation cycle started | Day 43
Pregnancy rates (per stimulation cycle and embryo transfer) | Throughout the study, estimate 1 year
Implantation rates | Throughout the study, estimate 1 year
Ongoing pregnancy rates (per stimulation cycle and embryo transfer) | Throughout the study, estimate 1 year
Clinical and biochemical miscarriages rates (per stimulation cycle and embryo transfer) | Throughout the study, estimate 1 year
Ectopic pregnancy rates (per stimulation cycle and embryo transfer) | Throughout the study, estimate 1 year
Live birth rates | Throughout the study, estimate 18 +/-3 months
Assessment and recording of adverse events | Throughout the study, estimate 18 +/-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Muñoz, Dr., Principal Investigator — Physician - Investigator
Locations (3):
- Spain (3):
  - IVI Alicante, Alicante, Valencia
  - IVI Madrid, Madrid
  - IVI Murcia, Murcia

IPD SHARING:
Plan to Share IPD: Undecided